CLINICAL TRIAL: NCT00002644
Title: International Breast Cancer Intervention Study: A Multicentre Trial of Tamoxifen to Prevent Breast Cancer
Brief Title: Tamoxifen for the Prevention of Breast Cancer in High-Risk Women
Acronym: IBIS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CDR0000064151; 2005-003091-38 (EudraCT Number); ISRCTN91879928 (Registry Identifier: ISRCTN)
Record Dates: First submitted 1999-11-01; First posted 2004-05-11 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; tamoxifen; prevention; IBIS
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamoxifen citrate (Experimental): Tamoxifen citrate 20 mg/day for 5 years
  Interventions: Drug: Tamoxifen Citrate 20Mg Tab
- Placebo (Placebo Comparator): Placebo 20 mg/day for 5 years
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tamoxifen Citrate 20Mg Tab — Tamoxifen Citrate 20Mg Tab
  Arms: Tamoxifen citrate
Other: Placebo — Placebo 20Mg Tab
  Arms: Placebo

SUMMARY:
The International Breast Cancer Intervention Study I (IBIS-I) was designed to investigate the use of tamoxifen in preventing breast cancer in women with a higher risk of developing the disease. Recruitment of women to IBIS-I ended in March 2001 and it recruited 7154 women from 36 centres in 9 countries. The results of the study showed that tamoxifen reduced the incidence of breast cancer by one third in these high risk women but with some serious side effects. IBIS-II was designed to continue the work started in IBIS-I by examining the role of anastrozole in the prevention of breast cancer which we hope will reduce breast cancer by even more than tamoxifen with less serious side effects.

DETAILED DESCRIPTION:
Established in 1992, the IBIS-I Study investigated the efficacy of tamoxifen (a hormonal drug used to prevent breast cancer) versus a placebo drug (taken daily for five years) in terms of reduction of breast cancer incidence in pre and postmenopausal women at high risk of developing breast cancer. It was a double-blind, randomised placebo-controlled trial that recruited 7,154 women internationally (of which 4,277 were UK participants), aged 35-70 years. The primary outcome measure was the incidence of breast cancer, including ductal carcinoma in situ (cancer cells in the lining of the breast milk duct) and side effects present in the patients were also investigated.

Recruitment to the study completed in 2001 and the intervention (placebo/tamoxifen) ended in 2007. In early 2008 the Research Ethics Committee (REC) approved the conversion of IBIS-I to an epidemiological cohort study. During 2007-2016 participants were followed-up via an annual postal questionnaire.

In 2002, initial results found that tamoxifen reduced the risk of invasive breast cancer by 31%. Mortality from non-breast cancer causes was not increased by tamoxifen. However, the analysis concluded that the overall risk/benefit ratio for the use of tamoxifen in prevention remained unclear and that continued follow-up of trial participants was essential. A 2007 analysis on long-term tamoxifen prophylaxis for breast cancer confirmed the preventive effect of tamoxifen in terms of breast cancer incidence and that this was constant for the entire follow-up period. No reduction in size of benefit was observed for up to ten years following participant randomisation. Additionally, tamoxifen-related side effects such as thrombo-embolism were not increased anymore after the 5-year treatment period. These results therefore demonstrate that the benefit-to-risk ratio of tamoxifen improves with increasing duration of follow-up. Thus, how much additional benefit will be seen long-term remains an important question.

ELIGIBILITY:
Inclusion criteria:

The entry criteria are based on a relative risk of at least two-fold for women aged 45-70 years, four-fold for women aged 40-44 years and ten-fold for women aged 35-39 years.

Age 45-70 years

1. First degree relative who developed breast cancer at age 50 or less
2. First degree relative who developed bilateral breast cancer
3. Two or more first or second degree relatives who developed breast cancer
4. Nulliparous and a first degree relative who developed breast cancer
5. Benign biopsy with proliferative disease and a first degree relative who developed breast cancer
6. Lobular carcinoma in situ
7. Atypical ductal or lobular hyperplasia in a benign lesion

19)Women at high risk who do not fit into the above categories (risk equivalent)*

* These women must have clearly apparent family history indicating at least two fold increased risk of breast cancer.

Age 40-44 years 8) Two or more first or second degree relatives who developed breast cancer at age 50 or less 9) First degree relative with bilateral breast cancer who developed the first breast cancer at age 50 or less 10) Nulliparous and a first degree relative who developed breast cancer at age 40 or less 11) Benign biopsy with proliferative disease and a first degree relative who developed breast cancer at age 40 or less 12) Lobular carcinoma in situ 13) Atypical ductal or lobular hyperplasia in a benign lesion 14) Women at high risk who do not fit into the above categories (risk equivalent)*

* These women must have clearly apparent family history indicating at least four fold increased risk of breast cancer.

Age 35-39 years 15) Two or more first degree relatives who developed breast cancer at age 50 or less 16) First degree relative with bilateral breast cancer who developed the first breast cancer at age 40 or less 17) Lobular carcinoma in situ 18) Women at high risk who do not fit into the above categories (risk equivalent)*

Exclusion criteria:

1. Pregnant, or at pregnancy risk. If necessary, pre and peri menopausal women must use non-hormonal contraception during the trial.
2. Any previous cancer (except non-melanoma skin cancer or in situ cancer of the cervix).
3. Life expectancy of less than 10 years or other medical condition more serious than the risk of breast cancer.
4. Psychologically and physically unsuitable for five years tamoxifen/placebo therapy.
5. Current treatment with anti-coagulants.
6. Previous deep vein thrombosis or pulmonary embolus.
7. Current tamoxifen use.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7154 (Actual)
Dates: Start 1994-01 (Actual); Primary Completion 2001-01 (Actual); Study Completion 2011-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Cuzick, PhD, Study Chair — Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, England, United Kingdom

REFERENCES:
- [Result] Cuzick J, Warwick J, Pinney E, Duffy SW, Cawthorn S, Howell A, Forbes JF, Warren RM. Tamoxifen-induced reduction in mammographic density and breast cancer risk reduction: a nested case-control study. J Natl Cancer Inst. 2011 May 4;103(9):744-52. doi: 10.1093/jnci/djr079. Epub 2011 Apr 11. PMID 21483019
- [Result] Stone J, Warren RM, Pinney E, Warwick J, Cuzick J. Determinants of percentage and area measures of mammographic density. Am J Epidemiol. 2009 Dec 15;170(12):1571-8. doi: 10.1093/aje/kwp313. Epub 2009 Nov 12. PMID 19910376
- [Result] Cuzick J, Forbes JF, Sestak I, Cawthorn S, Hamed H, Holli K, Howell A; International Breast Cancer Intervention Study I Investigators. Long-term results of tamoxifen prophylaxis for breast cancer--96-month follow-up of the randomized IBIS-I trial. J Natl Cancer Inst. 2007 Feb 21;99(4):272-82. doi: 10.1093/jnci/djk049. PMID 17312304
- [Result] Sestak I, Kealy R, Edwards R, Forbes J, Cuzick J. Influence of hormone replacement therapy on tamoxifen-induced vasomotor symptoms. J Clin Oncol. 2006 Aug 20;24(24):3991-6. doi: 10.1200/JCO.2005.04.3745. PMID 16921052
- [Result] Cuzick J, Warwick J, Pinney E, Warren RM, Duffy SW. Tamoxifen and breast density in women at increased risk of breast cancer. J Natl Cancer Inst. 2004 Apr 21;96(8):621-8. doi: 10.1093/jnci/djh106. PMID 15100340
- [Result] Cuzick J, Forbes J, Edwards R, Baum M, Cawthorn S, Coates A, Hamed A, Howell A, Powles T; IBIS investigators. First results from the International Breast Cancer Intervention Study (IBIS-I): a randomised prevention trial. Lancet. 2002 Sep 14;360(9336):817-24. doi: 10.1016/s0140-6736(02)09962-2. PMID 12243915
- [Result] Warwick J, Pinney E, Warren RM, Duffy SW, Howell A, Wilson M, Cuzick J. Breast density and breast cancer risk factors in a high-risk population. Breast. 2003 Feb;12(1):10-6. doi: 10.1016/s0960-9776(02)00212-6. PMID 14659350
- [Result] Sestak I, Kealy R, Nikoloff M, Fontecha M, Forbes JF, Howell A, Cuzick J. Relationships between CYP2D6 phenotype, breast cancer and hot flushes in women at high risk of breast cancer receiving prophylactic tamoxifen: results from the IBIS-I trial. Br J Cancer. 2012 Jul 10;107(2):230-3. doi: 10.1038/bjc.2012.278. Epub 2012 Jun 26. PMID 22735900
- [Result] Palva T, Ranta H, Koivisto AM, Pylkkanen L, Cuzick J, Holli K. A double-blind placebo-controlled study to evaluate endometrial safety and gynaecological symptoms in women treated for up to 5 years with tamoxifen or placebo - a substudy for IBIS I Breast Cancer Prevention Trial. Eur J Cancer. 2013 Jan;49(1):45-51. doi: 10.1016/j.ejca.2012.06.015. Epub 2012 Jul 23. PMID 22832202
- [Result] Cuzick J, Sestak I, Cawthorn S, Hamed H, Holli K, Howell A, Forbes JF; IBIS-I Investigators. Tamoxifen for prevention of breast cancer: extended long-term follow-up of the IBIS-I breast cancer prevention trial. Lancet Oncol. 2015 Jan;16(1):67-75. doi: 10.1016/S1470-2045(14)71171-4. Epub 2014 Dec 11. PMID 25497694
- [Result] Brentnall AR, Cuzick J, Byers H, Segal C, Reuter C, Detre S, Sestak I, Howell A, Powles TJ, Newman WG, Dowsett M. Relationship of ZNF423 and CTSO with breast cancer risk in two randomised tamoxifen prevention trials. Breast Cancer Res Treat. 2016 Aug;158(3):591-6. doi: 10.1007/s10549-016-3885-x. Epub 2016 Jul 11. PMID 27400912
- [Result] Cuzick J, Brentnall AR, Segal C, Byers H, Reuter C, Detre S, Lopez-Knowles E, Sestak I, Howell A, Powles TJ, Newman WG, Dowsett M. Impact of a Panel of 88 Single Nucleotide Polymorphisms on the Risk of Breast Cancer in High-Risk Women: Results From Two Randomized Tamoxifen Prevention Trials. J Clin Oncol. 2017 Mar;35(7):743-750. doi: 10.1200/JCO.2016.69.8944. Epub 2016 Dec 28. PMID 28029312
- [Result] Smith SG, Sestak I, Howell A, Forbes J, Cuzick J. Participant-Reported Symptoms and Their Effect on Long-Term Adherence in the International Breast Cancer Intervention Study I (IBIS I). J Clin Oncol. 2017 Aug 10;35(23):2666-2673. doi: 10.1200/JCO.2016.71.7439. Epub 2017 Jun 29. PMID 28661758